CLINICAL TRIAL: NCT01458327
Title: An Open-Label Proof-of-Principle Study Testing the Use of an Additional MDMA-Assisted Therapy Session in People Who Relapsed After Participating in a Phase 2 Clinical Trial of MDMA-Assisted Therapy to Treat Chronic, Treatment-Resistant Posttraumatic Stress Disorder
Brief Title: Additional MDMA-assisted Therapy for People Who Relapsed After MDMA-assisted Therapy Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP1-E2
Record Dates: First submitted 2011-10-12; First posted 2011-10-24 (Estimated); Results first posted 2021-11-03 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: MDMA; PTSD; therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDMA-assisted therapy (Experimental): One experimental session of MDMA-assisted therapy
  Interventions: Drug: Midomafetamine; Behavioral: Therapy

INTERVENTIONS:
Drug: Midomafetamine — 125 mg MDMA followed by 62.5 mg MDMA 1.5 to 2.5 hours later
  Other Names: MDMA; 3,4-methylenedioxymethamphetamine
Behavioral: Therapy — Non-directive therapy

SUMMARY:
This study will consist of a single session of MDMA-assisted therapy with a full dose of MDMA for people who took part in a study of MDMA-assisted therapy in people with posttraumatic stress disorder (PTSD) whose PTSD symptoms returned to higher levels at least a year after the first MDMA sessions. The single session will be performed by the same pair of therapists who performed the sessions in the first study. People will have a preparatory session, the MDMA-assisted session and three non-drug sessions afterward. Their PTSD symptoms and symptoms of depression will be measured at the start of this study and two and 12 months after the session.

DETAILED DESCRIPTION:
This study will investigate the effects of an additional 3,4-methylenedioxymethamine (MDMA)-assisted therapy session in up to three participants with PTSD who relapsed after their PTSD symptoms had significantly decreased during MAPS' initial U.S. Phase 2 trial testing the use of MDMA-assisted therapy in subjects with chronic, treatment-resistant posttraumatic stress disorder PTSD). This new protocol will consist of a single, full-dose open-label session of MDMA-assisted therapy, along with associated non-drug preparation and integrative therapy sessions.

MDMA is an investigational drug that was studied in a randomized, placebo-controlled study in 21 participants, and it included a final evaluation of symptoms at least one year after taking part in the study. While PTSD symptoms in most study subjects stayed at the same levels from when they completed the study, symptoms had returned in a few people. This open-label study is intended to see if an additional MDMA-assisted session conducted at least 14 months after the first sessions can help reduce PTSD symptoms.

The MDMA-assisted therapy session will be conducted by a male and female co-therapist team, one a psychiatrist and the other a psychiatric nurse. Vital signs (blood pressure, pulse and body temperature) and psychological distress will be measured throughout the experimental session. After the experimental session they will spend the night in the clinic with an attendant on duty, and complete a measure of alterations in consciousness, the States of Consciousness Questionnaire (SCQ) on the evening or day following the experimental session. Participants will meet with the investigators the next morning for an integrative therapy session before leaving the clinic. During integrative therapy sessions they will receive support in integrating their experiences and insights from the MDMA-assisted therapy session. There will be daily phone contact with one of the investigators for 7 days after the experimental session. Symptoms of PTSD, depression and general function will be assessed two months after the experimental session. There will be a long-term follow up with repeated outcome measures 12 months after the experimental session

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with chronic PTSD;
* Have a CAPS score showing moderate to severe PTSD symptoms;
* Have participated in MP-1;
* Are at least 18 years old;
* Must be generally healthy;
* Must sign a medical release for the investigators to communicate directly with their therapist and doctors;
* Are willing to refrain from taking any psychiatric medications during the study period;
* Willing to follow restrictions and guidelines concerning consumption of food, beverages, and nicotine the night before and just prior to each experimental session;
* Willing to remain overnight at the study site;
* Agree to have transportation other than driving themselves home or to where they are staying after the integrative session on the day after the MDMA session;
* Are willing to be contacted via telephone for all necessary telephone contacts;
* Must have a negative pregnancy test if able to bear children, and agree to use an effective form of birth control;
* must provide a contact in the event of a participant becoming suicidal;
* Are proficient in speaking and reading English;
* agree to have all clinic visit sessions recorded to audio and video
* Agree not to participate in any other interventional clinical trials during the duration of this study.

Exclusion Criteria:

* Are pregnant or nursing, or if a woman who can have children, those who are not practicing an effective means of birth control;
* Weigh less than 48 kg;
* Are abusing illegal drugs;
* Are unable to give adequate informed consent;
* Upon review of past and current drugs/medication must not be on or have taken a medication that is exclusionary;
* Upon review of medical or psychiatric history must not have any current or past diagnosis that would be considered a risk to participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-12-15 (Actual); Primary Completion 2014-06-27 (Actual); Study Completion 2014-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Mithoefer, MD, Principal Investigator — Psychiatrist
Locations (1):
- Offices of Michael Mithoefer, Mt. Pleasant, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 3,4-methylenedoxymethamphetamine (MDMA)-Assisted Therapy: 3,4-methylenedioxymethamphetmine (MDMA): 125 mg MDMA followed by 62.5 mg MDMA 1.5 to 2.5 hours later
  MDMA-AT: MDMA-assisted therapy
Period: Overall Study
Arm/Group | 3,4-methylenedoxymethamphetamine (MDMA)-Assisted Therapy
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 3,4-methylenedoxymethamphetamine (MDMA)-Assisted Therapy
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (7.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Baseline Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV)
Description: The CAPS-IV is a structured clinical interview designed to assess the symptoms and severity of PTSD. The CAPS-IV provides a means to evaluate the frequency and intensity dimensions of each symptom, the impact of symptoms on the patient's social and occupational functioning, the overall severity of the symptom complex, global improvement since baseline, and the validity of the ratings obtained. Total severity scores range from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: Less than 4 weeks before first experimental session
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 3,4-methylenedoxymethamphetamine (MDMA)-Assisted Therapy: 125 mg and 62.5 mg MDMA and therapy
  3,4-methylenedioxymethamphetmine (MDMA): 125 mg MDMA followed by 62.5 mg MDMA 1.5 to 2.5 hours later
  Therapy: MDMA-assisted therapy
Arm/Group | 3,4-methylenedoxymethamphetamine (MDMA)-Assisted Therapy
Number analyzed (Participants) | 3
score on a scale | 93.3 (1.53)

2. Primary Outcome: Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV) at 2-month Follow-up
Description: as for outcome 1
Time Frame: 2 months post experimental session
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3,4-methylenedoxymethamphetamine (MDMA)-Assisted Therapy
Number analyzed (Participants) | 3
score on a scale | 31.3 (12.01)

3. Primary Outcome: Clinician-Administered PTSD Scale (CAPS-IV)) at 12-month Follow-up
Description: The Clinician-Administered PTSD Scale for DSM-IV (CAPS-IV) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-IV. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.
Time Frame: 12 months post experimental session
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3,4-methylenedoxymethamphetamine (MDMA)-Assisted Therapy
Number analyzed (Participants) | 3
score on a scale | 52.7 (39.63)

4. Primary Outcome: Change in Clinician-Administered PTSD Scale (CAPS-IV) From Baseline to 2-month Follow-up
Description: as for outcome 3
Time Frame: Baseline to 2 months post experimental session
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3,4-methylenedoxymethamphetamine (MDMA)-Assisted Therapy
Number analyzed (Participants) | 3
score on a scale | -62.0 (12.53)

5. Primary Outcome: Change in Clinician-Administered PTSD Scale (CAPS-IV) From Baseline to 12-month Follow-up
Description: as for outcome 3
Time Frame: Baseline to 12 months post experimental session
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 3,4-methylenedoxymethamphetamine (MDMA)-Assisted Therapy
Number analyzed (Participants) | 3
score on a scale | -40.7 (40.27)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected throughout the study for approximately 12 months during Experimental Session (Visit 2), Integrative Sessions (Visit 3-5), 2-month Follow-up (Visit 6), and 12-month Follow-up (Visit7). AE's that occurred prior to date of first experimental dose were not reported.
Arm/Group | 3,4-methylenedoxymethamphetamine (MDMA)-Assisted Therapy
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3,4-methylenedoxymethamphetamine (MDMA)-Assisted Therapy (N=3)
Suicidal ideation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3,4-methylenedoxymethamphetamine (MDMA)-Assisted Therapy (N=3)
Major depression (Psychiatric disorders) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1)
Dissociation (Psychiatric disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2011-04-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT01458327/Prot_SAP_001.pdf
  • Informed Consent Form (2011-06-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT01458327/ICF_002.pdf